CLINICAL TRIAL: NCT04267354
Title: Arm Cycling in Facioscapulohumeral Dystrophy (FSHD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RL1 627
Record Dates: First submitted 2020-02-04; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm cycling (Experimental): Participants will perform arm cycling using a table-top arm cycler. Cadence and resistance of the exercise will be determined as per each individual's tolerance. All exercise will be supervised by the neuromuscular specialist physio, to ensure it is completed safely. Participants will be able to have plenty of breaks during the assessments.
  Interventions: Other: Arm cycling

INTERVENTIONS:
Other: Arm cycling — The arm cycle will be placed on table with height adjusted to be the same as the acromion (highest point on shoulder). Participants will start arm cycling at a low intensity and increase as per tolerance. They will exercise for a maximum of two minutes at a time, followed by a rest period for 30 seconds. In this manner 5 cycles of exercise and rest will be performed. The exercise sessions are anticipated to last a maximum of 20 minutes, depending on the patient's abilities.

SUMMARY:
The investigators believe that arm cycling has the potential to be effective in maintaining or improving shoulder muscle functioning. However, there is no evidence for its safety or effectiveness in the upper extremity. The aim of the study is to establish the ability of FSHD sufferers to perform arm cycling to underpin the future design of an arm exercise trial. The study hypothesis is that the limited range of shoulder movement and muscle weakness should not impact the ability of FSHD sufferers to perform arm cycling.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years
2. Genetically confirmed diagnosis of FSHD
3. Willing to attend the assessment session
4. Able to understand the participant information sheet and provide written informed consent

Exclusion Criteria:

1. Aged <18 years or >60 years
2. Co-morbidity that would affect their ability to perform arm cycling
3. Unwilling to complete the assessments of the study
4. Unable to understand the participant information sheet and provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | At one-off study visit: Prior to completion of exercise session
  A 12 item patient-reported shoulder instability questionnaire. Each of the questions presents five possible responses corresponding to a score of 0 (most disability/pain) to 4 (least disability/pain). when the twelve items are summed, the questionnaire then produces a single score with a range from 0 (most disability/pain) to 48 (least disability/pain).

SECONDARY OUTCOMES:
Range of movement | At one-off study visit: Prior to completion of exercise session
  A physiotherapist-assessed score of amount of movement at a joint in degrees, using goniometer. Range of movement is measured for both left and right shoulder joints in abduction, flexion and extension. Range of movement is measured for both left and right elbow joints in flexion and extension.
Strength of muscles at shoulder and elbow joints | At one-off study visit: Prior to completion of exercise session
  Assessment of muscle strength at at shoulder and elbow joints, by physiotherapist using a hand held dynamometer device. Using the dynamometer, the physiotherapist pushes against the joint and the patient resists. The dynamometer then provides a strength reading in Newton Metres of Torque. Both left and right shoulders will be assessed in abduction, flexion and extension. Both left and right elbows will be assessed in extension and flexion.
Resistance of arm cycling | At one-off study visit: During exercise session
  Patients will be asked to complete the arm cycling exercise at whatever resistance they feel most comfortable. Chosen resistance will be recorded.
Cadence of arm cycling | At one-off study visit: During exercise session
  Patients will be asked to complete the arm cycling exercise at whatever speed they feel most comfortable. The chosen cadence (speed) in cycles per minute will be recorded.
Borg Rate of Perceived Exertion (RPE) | At one-off study visit: During exercise session
  A patient-reported score of effort during exercise. The score ranges from 6 (no exertion at all) to 20 (maximal exertion). Patients will be asked to exercise at a level that is comfortable to them and indicate which RPE score they feel that they are working to, for each cycle of the arm cycling exercise.
Video analysis | At one-off study visit: During exercise session
  Video analysis of shoulder and elbow joint angles during arm cycling. Analysis software will be used to measure patient wrist, elbow and shoulder flexion and extension as well as trunk orientation during the exercise session.

OTHER OUTCOMES:
Patient suggestions | At one-off study visit: Immediately after completion of exercise session
  A free-text questionnaire asking patients to report any suggestions that they may have regarding factors that may limit their performance during this type of exercise, particularly if it were to be completed at home. There is no score for this question.
Patient willingness to continue | At one-off study visit: Immediately after completion of exercise session
  A free-text questionnaire asking patients to report whether they would be willing to continue with this sort of exercise at home, should it be proved effective. There is no score for this question.

CONTACTS AND LOCATIONS:
Overall Officials: Richa Kulshrestha, MBBS, MRCPCH, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No